CLINICAL TRIAL: NCT06563310
Title: Neurofeedback Enhanced Cognitive Reappraisal Training - Phase 4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stefanie Russman Block, Clinical Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HUM00209563 - phase 4; 1K23MH133063-01A1 (NIH)
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Social Anxiety Disorder; Panic Disorder; Generalized Anxiety Disorder
Keywords: functional magnetic resonance imaging
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Panic Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Veritable-NF (Experimental)
  Interventions: Other: Functional magnetic resonance imaging (fMRI) with Veritable-NF
- Sham-NF (Active Comparator)
  Interventions: Other: fMRI with Sham-NF

INTERVENTIONS:
Other: Functional magnetic resonance imaging (fMRI) with Veritable-NF — Participants will complete 4 visits (some can be done virtually). The baseline visit will include a clinical interview. Eligible participants will complete a series of questionnaires and a practice session at visit 2, and may do a mock scan if the visit is in person. Visit 3 will take place within 5 days of the practice session. Participants will have an fMRI with real neurofeedback and answer a series of questions pertaining to the scan. 2 weeks after visit 3, participants will revisit the questionnaires they completed at baseline. Visit 4 will take place one month after visit 3 and will include a follow-up interview with an assessor and the final questionnaire collection.
  Arms: Veritable-NF
Other: fMRI with Sham-NF — Participants will complete 4 visits (some can be done virtually). The baseline visit will include a clinical interview. Eligible participants will complete a series of questionnaires and a practice session at visit 2, and may do a mock scan if the visit is in person. Visit 3 will take place within 5 days of the practice session. Participants will have an fMRI with neurofeedback that looks similar to real neurofeedback but does not reflect their true brain signal. Afterwards, they will answer a series of questions pertaining to the scan. 2 weeks after visit 3, participants will revisit the questionnaires they completed at baseline. Visit 4 will take place one month after visit 3 and will include a follow-up interview with an assessor and the final questionnaire collection.
  Arms: Sham-NF

SUMMARY:
This study seeks to understand emotion regulation in those with young adults with anxiety using real-time functional magnetic resonance imaging neurofeedback, a tool that allows individuals to control brain activity. The goal of this project is to understand how receiving feedback about one's own brain activity relates to emotion regulation ability. This work will help the study team understand the brain areas involved in emotion regulation and could lay the groundwork to test if psychotherapy outcomes can be enhanced using neurofeedback.

The study hypotheses include:

* Participants receiving veritable-Neurofeedback (NF) will show a greater activation increases in the prefrontal cortex (PFC) compared to sham-NF
* Participants receiving veritable-NF will show greater cognitive reappraisal (CR) ability compared to those receiving sham-NF
* PFC activation will positively correlate with CR ability

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis (primary source of distress and/or interference) of generalized anxiety disorder, social anxiety disorder, panic disorder or illness anxiety disorder based on structured interview. Comorbid phobic disorders allowed, but these cannot be the primary source of interference or distress due to the lowered chances of encountering anxiety-provoking stimuli during the study period
* Score of 2 or more on at least 1 question from GAD/CROSS-AD composite
* Medically and physically able to consent
* Not regularly taking any medication, prescription or non-prescription, with psychotropic effects other than:

  1. Buspirone, or antidepressant (e.g., selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI)) with stable dosage for past 4 weeks
  2. The same oral hormonal contraceptive for at least 3 months
* For females, not currently pregnant or actively trying to become pregnant
* Ability to tolerate small, enclosed spaces without anxiety
* No metals, implants or metallic substances within or on the body that might cause adverse effects to the subject in a strong magnetic field, or interfere with image acquisition (per protocol)
* Size compatible with scanner gantry (per protocol)

Exclusion Criteria:

* Current diagnosis of Obsessive Compulsive Disorder, Posttraumatic Stress Disorder, or Bipolar Disorder
* Current substance abuse or dependence (past 6 months)
* Active suicidality with plan or intent
* Current psychosis
* History of serious neurological illness or current medical condition that could compromise brain function, such as liver failure
* History of closed head injury, e.g., loss of consciousness greater (>) approximately (~) 5 minutes, hospitalization, neurological sequela

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Change in prefrontal cortex (PFC) activity (baseline to transfer run) from the reappraise > look contrast | Approximately 60 minutes
Change in negative affect ratings of images from the International Affective Picture System (IAPS) | Approximately 60 minutes
  The Self-Assessment Manikin (SAM) is a pictorial assessment technique in which a changing manikin figure depicts values along the primary dimension of affective valence (positive/negative). Users may indicate emotional reactions along a scale from 1-9, with higher numbers indicating greater negative affect. After the scan, participants will rate each image they saw from the IAPS along this scale. Differences in SAM ratings from look to reappraise trials will be evaluated and compared between sham-NF and veritable-NF groups.

SECONDARY OUTCOMES:
Change in amygdala-PFC functional connectivity (baseline to transfer) from reappraise > look contrast | Approximately 60 minutes
  To examine amygdala connectivity, the study team will use a psychophysiological interaction analysis. Deconvolved time series from anatomical left and right amygdala seeds for each participant will be multiplied by a vector for the reappraise > look contrast at each run (baseline, Neruofeedback1 (NF1), NF2, NF3, transfer). Regressors for the seed time series, the original condition and the interaction term will be convolved with the canonical hemodynamic response function. Change in connectivity from pre-to-post training will be calculated by subtracting the baseline-run contrast map from the transfer-run contrast map. Resulting contrast maps will be entered into second-level random effects analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Russman Block, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No